CLINICAL TRIAL: NCT06483945
Title: Dexcom Continuous Glucose Monitoring System Use in aReal-World, Global Registry
Brief Title: Dexcom Continuous Glucose Monitoring System Use in aReal-World, Global Registry (Dexcom Global Registry)
Status: Recruiting | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-1000088
Record Dates: First submitted 2024-03-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Dexcom CGM G6/G6 Pro/G7 — Dexcom CGM G6/G6 Pro/G7 device

SUMMARY:
"To evaluate the use of the Dexcom CGM System when used according to approved commercial labeling during standard clinical use and its impact on intended users in a real-world setting"

DETAILED DESCRIPTION:
"The Dexcom Global Registry is a non-randomized, open-label, multi-center registry with the goal of collecting Dexcom CGM System data in a real world setting.The registry study involves retrospective and/or prospective data collection associated with Dexcom CGM System use."

ELIGIBILITY:
Inclusion Criteria:

* Meets Dexcom CGM System Indications for Use (IFU) per approved commercial labeling
* Has at least one HbA1C (Hemoglobin a1c) measurement within three (3) months prior to the Dexcom CGM System use start date that is at least three (3) months after any prior CGM use
* Subject is willing and able to use Dexcom CGM System according to approved product labeling
* Subject is willing and able to complete applicable patient reported outcome assessments/ surveys
* Subject is willing and able to comply with the protocol
* Subject is willing and able to comply with provider requirements for at least two provider encounters per year according to applicable clinical practice guidelines
* Subject or the subject's legally authorized representative must provide written informed consent prior to any study-related data collection or be enrolled under an IRB/EC approved waiver of consent

Exclusion Criteria:

* Is contraindicated for a Dexcom CGM System per approved commercial labeling
* In the Investigator's opinion, the subject is not considered to be a suitable candidate

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The clinical study population will consist of up to 5000 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes (PROs) | 4 years
  Patients will be asked to complete multiple questionnaires over a period of 4 years for data to be analyzed and reported.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute of Endocrinology Diabetes, Health & Hormones, Stockbridge, Georgia
  - Palm Research Center, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No